CLINICAL TRIAL: NCT06479382
Title: A Prospective Early-Feasibility Study to Evaluate the Safety and Effectiveness of ETX-4143 2.0 Device in Subjects With Eye Pain
Brief Title: Study of the ETX-4143 2.0 Device in Subjects With Eye Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeCool Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETX4143-A002
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Eye Pain
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational (Experimental): Treatment with the ETX-4143 2.0 device
  Interventions: Device: ETX-4143 2.0
- Control (Sham Comparator): Treatment with a sham ETX-4143 2.0 device
  Interventions: Device: ETX-4143 2.0

INTERVENTIONS:
Device: ETX-4143 2.0 — Treatment of the eye with the ETX-4143 2.0 device

SUMMARY:
A prospective early-feasibility study to evaluate the safety and effectiveness of the ETX-4143 2.0 device. The device is intended to treat subjects with eye pain

DETAILED DESCRIPTION:
A prospective early-feasibility study to evaluate the safety and effectiveness of the ETX-4143 2.0 device. The device is intended to treat subjects who suffer from eye pain an do not get relieve from current medications or clinical treatments. Thirty eyes will be enrolled and randomized 2:1 to the investigational treatment or a sham treatment. Improvement in self-reported ocular pain and clinical safety measures will be evaluated.

It is anticipated that the learnings from the study will be used to design future study of the ETX-4143 2.0 device.

All subjects will be followed for 8 weeks. Subjects will only have the worse eye treated if both eyes meet the inclusion/exclusion criteria.

A medical monitor will evaluate the safety of the study on a continual basis.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of eye pain with no relief from currently available medications or treatments
* Willing to forgo participation in any other clinical stud for the duration of this study
* Demonstrate sufficient cognitive awareness to comply with the examination process
* Willing and able to comply with the schedule for follow-up visits
* Willing to participate in the study as evidenced by signing an informed consent document

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study time period, including the follow-up period
* Any active ocular infection or active ocular inflammation at the time of the screening visit
* History of herpes keratitis, non-healing corneal epithelial defects, or neurotrophic keratopathy due to corneal herpetic disease, stem cell deficiency, diabetic keratopathy, severe lagophthalmos, or topical anesthetic abuse
* Any history of significant eye surgery with the prior 90 days
* Planned eye surgery during the entire study
* Participation in any clinical study of an investigational product within 30 days prior to enrollment
* Any history of serious, poorly controlled systemic or ophthalmic condition that could compromise the subject's ability to comply with the protocol or compromise their safety

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Reduction of eye pain | Eight weeks
  Patient reported level of eye pain
Adverse events | Eight weeks
  Adverse events related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Casey, OD, Study Chair — VP of Clinical Develpment
Locations (4):
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Ophthamic Trials Australia, Brisbane, Queensland
  - Innovative Eye Care, Adelaide, South Australia
  - Sunshine Eye Surgeons, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: No